CLINICAL TRIAL: NCT02335788
Title: EMBA Peripheral Embolization Device ("EPED") Study
Acronym: EPED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EMBA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRT-EPE-0028
Record Dates: First submitted 2015-01-06; First posted 2015-01-12 (Estimated); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Peripheral Embolization
Keywords: Therapeutic; Embolization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm - EMBA PED (Other): The EMBA Peripheral Embolization Device when indicated for arterial and venous embolization in the peripheral vasculature.
  Interventions: Device: The EMBA Peripheral Embolization Device

INTERVENTIONS:
Device: The EMBA Peripheral Embolization Device — arterial and venous embolization in the peripheral vasculature

SUMMARY:
This is an open label, acute, non-randomized, prospective, "first in man" (FIM) single-center study of the EMBA Medical Peripheral Embolization Device (PED).

DETAILED DESCRIPTION:
This study is a FIM, open label, prospective, single center, non-randomized, evaluation of the EMBA Medical Peripheral Embolization Device (PED) used for arterial or venous embolization in the peripheral vasculature.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is >18 years of age.
2. Patient is considered a candidate for arterial or venous embolization in the peripheral vasculature.
3. Patient has a target vessel diameter of 3-8mm and a target PED landing zone of greater than 25mm wherein the vessel diameter is between 3 and 8 mm.
4. The patient or legal guardian has been informed of the nature of the study and agrees to its provisions and has provided informed written consent.
5. The patient has suitable vessel anatomy that would allow proper placement of the PED.

Exclusion Criteria:

1. The patient has one of the following conditions:

   1.1 Arterio-venous fistula 1.2 Hypercoagulability 1.3 Systemic coagulopathy 1.4 Connective tissue disorder such as Ehlers-Danlos Syndrome 1.5 Congenital arteritis such as Takayasu's Disease 1.6 Other circulatory disorders at the discretion of the implanting physician
2. The patient has an uncontrolled infectious disease.
3. The patient has a life expectancy of less than 6 months.
4. The patient is pregnant.
5. The patient has a condition that inhibits radiographic visualization of the PED.
6. The patient has a known allergy or intolerance to Nitinol.
7. The patient has a known hypersensitivity to contrast that cannot be pre-treated.
8. The patient's access vessels preclude safe insertion of the delivery system.
9. The patient is currently participating in another device or drug study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Target vessel occlusion (assessed by CTA) | 30 Days
  vessel occlusion as assessed by CTA

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Holden, MD, Principal Investigator — Auckland City Hospital
Locations (1):
- Auckland City Hospital, Grafton, Auckland, New Zealand